CLINICAL TRIAL: NCT00267241
Title: Effects of Different Assisted Mechanical Ventilation in ALI/ARDS Patients
Brief Title: Effects of Different Assisted Mechanical Ventilation in Acute Lung Injury (ALI)/Acute Respiratory Distress Syndrome (ARDS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1600
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: ARDS; ALI; respiratory mechanics; gas exchange; assisted ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ALI/ARDS patients
  Interventions: Other: Mechanical Ventilation

INTERVENTIONS:
Other: Mechanical Ventilation — Four different types of assisted ventilation (pressure support, pressure support plus sigh, BIPAP, variable ventilation)

SUMMARY:
The aim of this study is to evaluate the effects in terms of gas exchange, respiratory mechanics and comfort of breathing, of different assisted mechanical ventilation in ALI/ARDS patients.

DETAILED DESCRIPTION:
ALI/ARDS patients (during assisted ventilation) will be ventilated with different types of assisted ventilation (pressure support, pressure support plus sigh, BIPAP, variable ventilation) and gas exchange, comfort of breathing, respiratory mechanics and pattern of breathing will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALI/ARDS

Exclusion Criteria:

* COPD patients
* Barotrauma
* Hemodynamic instability
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Gas exchange and respiratory mechanics | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy